CLINICAL TRIAL: NCT02794727
Title: Physical Activity in the Medical Workplace- a Way to Improve Physical and Mental Well-being?
Brief Title: Physical Activity in the Medical Workplace
Acronym: OPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ivana Croghan, PhD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-003049
Record Dates: First submitted 2016-06-02; First posted 2016-06-09 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blinded Fitbit (Sham Comparator): Subjects will wear the physical activity monitor (fitbit) for 12 weeks but will be blinded to the monitor display.
  Interventions: Device: Blinded Fitbit
- Unblinded Fitbit (Active Comparator): Subjects will wear the physical activity monitor (fitbit) for 12 weeks. They will have access to the monitor display and will have consults with study physician to set goals for the duration of the study.
  Interventions: Device: Unblinded Fitbit
- No Fitbit (No Intervention): Subjects will not wear any activity monitor for 12 weeks.

INTERVENTIONS:
Device: Blinded Fitbit — Subjects will wear a blinded Fitbit to monitor activity while in the workplace for 12 weeks.
  Arms: Blinded Fitbit
Device: Unblinded Fitbit — Subjects will be unblinded to the Fitbit display for 12 weeks with set activity goals.
  Arms: Unblinded Fitbit

SUMMARY:
Decreased physical activity is not only associated with multiple chronic medical conditions, including obesity, but also with depressed mood, and other negative emotions. As many employed adults spend a great deal of time at work where we are predominantly sedentary, strategies to increase physical activity at work are being pursued to help improve the physical and mental health of Americans. This 17 week randomized controlled trial will investigate changes of occupational physical activity in three groups: those provided with a FitBit® but not able to monitor their activity level, and those provided with activity goals and individual physical activity challenges, and those who do not use a FitBit®.

DETAILED DESCRIPTION:
All subjects will be entered into a 4 week run-in phase where subjects will wear a blinded Fitbit during work hours. The baseline work activity is collected at this time. This phase is followed by a randomization to one of 3 groups: the blinded Fitbit group, the unblinded Fitbit group, and the group which will not wear any activity monitors. During these 12 weeks we will collect data on activity levels during work hours. Everyone will have a final contact at week 17 to close out the study.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 - 65 years of age
* Be a Mayo Clinic employee at 0.75 FTE or more
* Have no previous use of any activity monitor for 14 consecutive days or more
* Not be pregnant by subject self report
* Have a stable weight - defined as self-reported weight that has not changed more than 10% in the past 3 months
* Not have any previous history of joint problems that limit free movement, as determined by the PI
* Be able to participate fully in all aspects of the study
* Have understood and signed study informed consent.

Exclusion Criteria:

* Have a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence or skew data collection - such as a position where they predominantly provide transport as part of their job.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-06; Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T Croghan, PhD, Study Chair — Mayo Cinic; Ryan T Hurt, MD, PhD, Study Director — Mayo Clinic; Sanjeev Nanda, MD, Principal Investigator — Mayo Clinic; Sara Bonnes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nanda S, Hurt RT, Croghan IT, Mundi MS, Gifford SL, Schroeder DR, Fischer KM, Bonnes SL. Improving Physical Activity and Body Composition in a Medical Workplace Using Brief Goal Setting. Mayo Clin Proc Innov Qual Outcomes. 2019 Oct 16;3(4):495-505. doi: 10.1016/j.mayocpiqo.2019.07.002. eCollection 2019 Dec. PMID 31993569
- See also: pub med link to published study data — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6978599/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blinded Fitbit | Unblinded Fitbit | No Fitbit
Started | 44 | 46 | 45
Completed | 44 | 46 | 44
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinded Fitbit | Unblinded Fitbit | No Fitbit | Total
Number analyzed (Participants) | 44 | 46 | 45 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 46 | 45 | 135
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.3) | 40.4 (9.7) | 45.5 (9.8) | 42.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 39 | 114
  Male | 7 | 8 | 6 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white, non-hispanic | 38 | 42 | 43 | 123
  other | 6 | 4 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Fitbit Step Count Per Day
Description: change in number of daily steps as measured by the fitbit monitor
Time Frame: Baseline through Week 16
Measure: Least Squares Mean (Standard Error); unit: steps
Arm/Group | Blinded Fitbit | Unblinded Fitbit
Number analyzed (Participants) | 44 | 46
steps | -323.5 (90.5) | 321.2 (88.4)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Blinded Fitbit | Unblinded Fitbit | No Fitbit
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46 | 1/45
Other Adverse Events (participants affected / at risk) | 6/44 | 4/46 | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Fitbit (N=44) | Unblinded Fitbit (N=46) | No Fitbit (N=45)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Hospitalization due to unprovoked pulmonary embolism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Fitbit (N=44) | Unblinded Fitbit (N=46) | No Fitbit (N=45)
musculoskeletal pain/trauma (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
dental implant/root canal (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
foot nerve pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
ear/sinus infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
GI pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT02794727/Prot_SAP_000.pdf